CLINICAL TRIAL: NCT07332377
Title: PsyMINT: Mobile Health (mHealth) Intervention to Support Self-Management of Pain and Symptoms for Cancer Survivors
Brief Title: mHealth Intervention for Pain Self Management
Acronym: PsyMINT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-25-22625; HM300000094 (Other: Virginia Commonwealth University); P50MD017319 (NIH)
Record Dates: First submitted 2026-01-08; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pain; Pain Management; Symptom Monitoring; Symptom Management; Cancer Survivorship
Keywords: cancer survivorship; pain management; mHealth; behavioral intervention; nonpharmacologic intervention; app; digital health
MeSH Terms: conditions — Pain; Agnosia; Alzheimer Disease | interventions — Telemedicine; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile Health (mHealth) Intervention (Experimental): Implement a bank of 60 mHealth intervention messages, ecological momentary assessments (EMAs), and e-diary entries to PiLR to deliver a 1-week mHealth intervention to cancer survivors experiencing pain
  Interventions: Behavioral: Mobile Health (mHealth) Intervention

INTERVENTIONS:
Behavioral: Mobile Health (mHealth) Intervention — Individuals will use the mHealth app for 1 week. Participants will interact with evidence-based messages and will complete ecological momentary assessments (EMA's) (two times per day) and electronic diaries (e-diaries) daily.

SUMMARY:
This is a feasibility pilot test of a single-arm intervention to evaluate the beta version of an mHealth app-based behavioral intervention prior to scaling for a randomized controlled trial (RCT). This mHealth intervention is designed to enhance self-efficacy and support pain and symptom self-management among post-treatment cancer survivors.

DETAILED DESCRIPTION:
The intervention involves a set of tested intervention messages, ecological momentary assessments (EMAs), and e-diary entries to our PsyMINT mobile app. A 1-week mHealth intervention to cancer survivors who experience pain will be delivered. The feasibility of an mHealth app platform (PsyMINT) as a message presentation environment will be delivered and evaluated. The app messages will target five topics/modules, including psychoeducational materials related to pain management; positive psychology; opioid literacy; skill building for patient-provider communication and trust; and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* In a post-treatment stage with no evidence of disease (complete remission)
* Diagnosed with cancer in the past three years
* Experiencing cancer/treatment-related pain
* ≥ 18 years of age at the time of first diagnosis
* Cognitively able to actively participate in an online-based study
* Able to read, write, and understand English

Exclusion Criteria:

* Individuals who currently use any medication for psychiatric reasons (including stimulants, and mood stabilizers)
* Patients with major psychotic disorders (bipolar disorder or schizophrenia) and/or substance use disorders.
* Those who are currently pregnant or plan to become pregnant in the next three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of the mobile health (mHealth) intervention | Baseline and end of one week intervention
  The feasibility and acceptability of the behavioral intervention will be assessed using a pre-validated measure, the 19-item Post-Study System Usability Questionnaire (PSSUQ)87 (e.g., "It was simple to use this app") on a 7-point Likert scale. Acceptability and feasibility outcomes will be evaluated through analysis of mean scores and proportions, including:
  * Proportion of participants retained,
  * Proportion who complete at least 80% of EMAs,
  * 19-item Post-Study System Usability Questionnaire (PSSUQ) mean scores to be greater than 5 (as indicators of feasibility and acceptability).

SECONDARY OUTCOMES:
Self-efficacy for pain management | Baseline and end of one week intervention
  Determine preliminary evidence for efficacy, using the 10-item Pain Self-Efficacy Questionnaire (PSEQ) at baseline and at post-intervention.
Improved quality of life using a brief version of the Functional Assessment of Cancer Therapy (FACT-G) | Baseline and end of one week intervention
  Determine preliminary evidence of efficacy using a modified version (shortened) of the Functional Assessment of Cancer Therapy (FACT-G) at baseline and post-intervention. The 26-item FACT-G questionnaire is designed to assess 4 domains of health related quality of life in cancer patients: Physical, social, emotional, and functional well-being using a 5-point Likert scale (1 = Not at all through 5=Very much).
  For the FACT-G questionnaire, difference scores will be calculated for the four subscales and the total score using measurements obtained at baseline and post-intervention. The scoring is designed so that a lower score reflects an improved state of well-being and functioning.
Improved Quality of Life using the European Organization for Research and Treatment of Cancer (EORTC)'s Quality of Life Questionnaire (QLQ-C30) | Baseline and end of one week intervention
  Determine preliminary evidence of efficacy using the European Organization for Research and Treatment of Cancer (EORTC)'s Quality of Life Questionnaire (QLQ-C30) at baseline and at post-intervention. The 30-item EORTC is designed to measure health-related quality of life, including global health status, functional domains (physical, role, emotional, cognitive, and social functioning), and common cancer-related symptoms. We will compute mean scores of these sub-domains which will be reported on a 4 point Likert scale (1= Not at all 4 = Very much). Mean scores for global health status, symptom scales, and functional scales will be computed for measurements assessed at baseline and post-intervention, and difference scores for each subscale will be calculated. Low scores indicate better functioning and improved symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sun Jung Kim, Ph.D, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual data, but a de-identified aggregated form of self-report data may be available to share when the study is complete and findings are published.